CLINICAL TRIAL: NCT00740701
Title: fMRI and TMS Analysis of Cerebellar Cognitive Function
Brief Title: Effects of Transcranial Magnetic Stimulation to the Cerebellum on Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NA_00044841; R01MH060234 (NIH)
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Cognitive Performance
Keywords: TMS; fMRI; verbal working memory; classical conditioning; eyeblink; classical eyeblink conditioning; Healthy subjects; Memory

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham TMS (Sham Comparator): A Sham TMS coil, designed to elicit sham cerebellar transcranial magnetic stimulation, is used to administer sham TMS pulses after letters are presented.
  Interventions: Device: Cerebellar transcranial magnetic stimulation
- TMS (Experimental): A genuine TMS coil is used to administer cerebellar transcranial magnetic stimulation pulses after letter presentation.
  Interventions: Device: Cerebellar transcranial magnetic stimulation

INTERVENTIONS:
Device: Cerebellar transcranial magnetic stimulation — single pulse TMS or repetitive TMS at 1 Hz frequency

SUMMARY:
Functional neuroimaging studies have shown that the cerebellum is active during cognitive performance. The investigators hypothesize that stimulation of the cerebellum with transcranial magnetic stimulation will produce brief changes in performance of the task, suggesting that cerebellar activation is necessary for normal cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* 19-30 years of age
* Informed consent

Exclusion Criteria:

* History of seizure or a family history of epilepsy
* History of stroke
* Presence of metal anywhere in the head except the mouth
* Presence of cardiac pacemakers
* Presence of cochlear implants
* Presence of implanted medication pump
* History of heart disease
* Presence of intracardiac lines
* Increased intracranial pressure, such as after infarctions or trauma
* Children, or outside of age range
* Pregnancy
* Currently taking tricyclic anti-depressants or neuroleptic medication
* History of head trauma
* History of respiratory disease

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2000-04; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Behavioral performance (accuracy, or rate of conditioned responses) | during computerized task performance (2 hours)

SECONDARY OUTCOMES:
Reaction time | during performance of computerized task (2 hours)

CONTACTS AND LOCATIONS:
Overall Officials: John E Desmond, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States